CLINICAL TRIAL: NCT00567879
Title: A Phase Ib/IIa Trial of Panobinostat in Combination With Trastuzumab in Adult Female Patients With HER2 Positive Metastatic Breast Cancer Whose Disease Has Progressed During or Following Therapy With Trastuzumab
Brief Title: A Trial of Panobinostat and Trastuzumab for Adult Female Patients With HER2 Positive Metastatic Breast Cancer (MBC) Whose Disease Has Progressed on or After Trastuzumab
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to insufficient evidence of clinical benefit.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589C2204; 2007-002449-19 (EudraCT Number)
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HER2 positive; adult-female; LBH589; HDAC inhibitor; panobinostat
MeSH Terms: conditions — Breast Neoplasms | interventions — Panobinostat; Trastuzumab

ARMS (1):
- Panobinostat with trastuzumab (Experimental): Panobinostat intravenously (i.v.) or orally was given in combination with trastuzumab.
  Interventions: Drug: Panobinostat; Drug: Trastuzumab

INTERVENTIONS:
Drug: Panobinostat — Participants received escalating doses of panobinostat until the maximum tolerated dose (MTD) was reached. The starting dose of panobinostat i.v. was 10mg/m^2 at days 1 and 8 during a 21-day treatment cycle. The oral panobinostat starting dose was 20 mg twice weekly.
Drug: Trastuzumab — Fixed doses of trastuzumab were given in parallel with panobinostat. Trastuzumab i.v. was given weekly according to the instruction in the package insert.
  Other Names: Herceptin

SUMMARY:
The primary purpose of this study is to identify the maximum tolerated dose (MTD) of both intravenous and oral panobinostat plus trastuzumab. The study will evaluate safety and efficacy of the combination in adult female patients with HER2+ metastatic breast cancer

DETAILED DESCRIPTION:
This phase Ib/IIa study was prematurely terminated due to lack of efficacy noted in 55 patients with HER2-positive MBC who had progressed on or following a trastuzumab-based therapy.

ELIGIBILITY:
Key Inclusion criteria:

* Age > 18 year old
* Confirmed HER2+ ve metastatic breast cancer
* Prior treatment and progression on trastuzumab
* Patients must have adequate laboratory values
* Eastern Cooperative Oncology Group (ECOG) performance status of <2

Key Exclusion criteria:

* Patients with active central nervous system (CNS) disease or brain metastases except those who have been previously treated and have been stable for at least 3 months.
* Impaired heart function or clinically significant heart disease
* Impairment of gastrointestinal (GI) function, or GI disease that may significantly alter the absorption of LBH589
* Ongoing diarrhea
* Liver or renal disease with impaired hepatic or renal functions
* Concomitant use of any anti-cancer therapy or certain drugs
* Female patients who are pregnant or breast feeding
* Patients not willing to use an effective method of birth control

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- United States (7):
  - University of California at Los Angeles, Los Angeles, California
  - University of Colorado Dept. of Univ. of Colorado, Aurora, Colorado
  - Norwalk Hospital Dept of Norwalk Hospital (2), Norwalk, Connecticut
  - VA Maryland Health Care Dept.of GreenbaumCancerCent(3), Baltimore, Maryland
  - The Center for Cancer Care and Research, St Louis, Missouri
  - Ohio State Comprehensive Cancer Center/James Cancer Hospital SC, Columbus, Ohio
  - University of Pittsburgh Cancer Institute Dept of Magee Women's Hospital, Pittsburgh, Pennsylvania
- Canada (3):
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (3):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain Cédex
- Novartis Investigative Site, Heidelberg, Germany
- Italy (3):
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Modena, MO
- United Kingdom (3):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were allocated to dose escalation arm 1 (i.v. panobinostat) or arm 2 (oral panobinostat) according to a pre-determined sequence in the ratio 1:1. Each cohort consisted of newly enrolled participants. This study included a dose escalation phase to establish the maximum tolerated dose (MTD) and a dose expansion phase.
Groups:
- Escalation: i.v. Arm - 10mg/m^2: 10 mg/m^2 i.v. was given on day 1 and day 8 of a 21 day cycle.
- Escalation: i.v. Arm - 15mg/m^2: 15 mg/m^2 i.v. was given on day 1 and day 8 of a 21 day cycle.
- Escalation/Expansion: i.v. Arm -20mg/m^2: 20 mg/m^2 i.v. was given on day 1 and day 8 of a 21 day cycle.
- Oral Arm - Schedule A 20mg: 20 mg was given twice weekly for two consecutive weeks as part of a 21-day treatment cycle.
- Oral Arm - Schedule B 15 mg: 15 mg was given three times weekly for two consecutive weeks as part of a 21-day treatment cycle.
- Oral Arm - Schedule B 20mg: 20 mg was given three times weekly for two consecutive weeks as part of a 21-day treatment cycle.
Period: Overall Study
Arm/Group | Escalation: i.v. Arm - 10mg/m^2 | Escalation: i.v. Arm - 15mg/m^2 | Escalation/Expansion: i.v. Arm -20mg/m^2 | Oral Arm - Schedule A 20mg | Oral Arm - Schedule B 15 mg | Oral Arm - Schedule B 20mg
Started | 7 | 7 | 21 (7 participants belonged to the dose expansion group at 20mg/m2 i.v.) | 6 | 12 | 3
Maximum Tolerated Dose Determining Set | 5 | 7 | 18 (6 participants belonged to the dose expansion group at 20mg/m2 i.v.) | 6 | 12 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 7 | 21 | 6 | 12 | 3
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 1 | 0
Not completed — Abnormal test procedure(s) | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 0 | 0
Not completed — New cancer therapy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Disease progression | 5 | 7 | 15 | 5 | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Oral Arm - Schedule B 15mg: 15 mg was given three times weekly for two consecutive weeks as part of a 21-day treatment cycle.
- Total: Total of all reporting groups
Arm/Group | Escalation: i.v. Arm - 10mg/m^2 | Escalation: i.v. Arm - 15mg/m^2 | Escalation/Expansion: i.v. Arm -20mg/m^2 | Oral Arm - Schedule A 20mg | Oral Arm - Schedule B 15mg | Oral Arm - Schedule B 20mg | Total
Number analyzed (Participants) | 7 | 7 | 21 | 6 | 12 | 3 | 56
Age, Continuous [Median (Full Range); unit: Years] | 58.0 [35.0 to 60.0] | 49.0 [33.0 to 60.0] | 57.0 [37.0 to 83.0] | 54.5 [49.0 to 59.0] | 53.5 [40.0 to 65.0] | 47.0 [38.0 to 60.0] | 53.0 [33.0 to 83.0]
Sex/Gender, Customized [Number; unit: Participants]
  Female | 7 | 7 | 21 | 6 | 12 | 3 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Safety data was reviewed to determine the DLTs. DLTs comprised adverse events (AEs) or abnormal laboratory values that occurred at any time and were assessed as clinically relevant and meeting any of the following criteria: considered to be related to the study treatment and unrelated to disease, disease progression, inter-current illness, or concomitant medications. Toxicities were assessed using the National Cancer Institute common terminology criteria for adverse events (NCI CTCAE), version 3.0. Disease related symptoms were not considered a DLT.
Time Frame: day 21
Population: The Maximum Tolerated Dose (MTD) determining set was used for this analysis. The MTD determining set consisted of all participants who either received sufficient study drug and had sufficient safety evaluations or discontinued due to unacceptable toxicity.
Measure: Number; unit: Participants
Groups:
- Expansion: i.v. Arm -20mg/m^2: 20 mg/m^2 i.v. was given on day 1 and day 8 of a 21 day cycle.
Arm/Group | Escalation: i.v. Arm - 10mg/m^2 | Escalation: i.v. Arm - 15mg/m^2 | Escalation/Expansion: i.v. Arm -20mg/m^2 | Expansion: i.v. Arm -20mg/m^2 | Oral Arm - Schedule A 20mg | Oral Arm - Schedule B 15 mg | Oral Arm - Schedule B 20mg
Number analyzed (Participants) | 5 | 7 | 12 | 6 | 6 | 12 | 3
Participants | 0 | 0 | 1 | 1 | 1 | 3 | 1

2. Secondary Outcome: Number of Participants With Best Overall Response
Description: Tumors were assessed according to Response Evaluation Criteria in Solid tumors (RECIST). Complete response (CR): disappearance of all lesions (i.e. all evidence of disease, not just the target lesions) determined by 2 observations not less than 4 weeks apart; Partial response (PR): > 30% decrease in the sum of longest diameters of target lesions compared to baseline, with response or stable disease observed in non-target lesions, and no new lesions; Stable disease (SD): neither sufficient shrinkage to qualify for response or sufficient increase to qualify for progressive disease in target lesions, with response or stable disease observed in non-target lesions, and no new lesions; Progressive disease (PD): > 20% increase in the sum of longest diameters of target lesions compared to smallest sum longest diameter recorded. In addition, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: day 21
Population: The full analysis set was analyzed. The full analysis set included all randomized participants.
Measure: Number; unit: Participants
Arm/Group | Escalation: i.v. Arm - 10mg/m^2 | Escalation: i.v. Arm - 15mg/m^2 | Escalation/Expansion: i.v. Arm -20mg/m^2 | Oral Arm - Schedule A 20mg | Oral Arm - Schedule B 15 mg | Oral Arm - Schedule B 20mg
Number analyzed (Participants) | 7 | 7 | 21 | 6 | 12 | 3
Participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 1 | 0 | 0 | 0
  Stable disease | 4 | 1 | 8 | 1 | 3 | 0
  Progressive disease | 3 | 6 | 9 | 4 | 7 | 3
  Unknown | 0 | 0 | 3 | 1 | 2 | 0

ADVERSE EVENTS:
Arm/Group | Escalation: i.v. Arm - 10mg/m^2 | Escalation: i.v. Arm - 15mg/m^2 | Escalation/Expansion: i.v. Arm -20mg/m^2 | Oral Arm - Schedule A 20mg | Oral Arm - Schedule B 15 mg | Oral Arm - Schedule B 20mg
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/7 | 5/21 | 3/6 | 2/12 | 1/3
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 21/21 | 6/6 | 12/12 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation: i.v. Arm - 10mg/m^2 (N=7) | Escalation: i.v. Arm - 15mg/m^2 (N=7) | Escalation/Expansion: i.v. Arm -20mg/m^2 (N=21) | Oral Arm - Schedule A 20mg (N=6) | Oral Arm - Schedule B 15 mg (N=12) | Oral Arm - Schedule B 20mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic duct obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escalation: i.v. Arm - 10mg/m^2 (N=7) | Escalation: i.v. Arm - 15mg/m^2 (N=7) | Escalation/Expansion: i.v. Arm -20mg/m^2 (N=21) | Oral Arm - Schedule A 20mg (N=6) | Oral Arm - Schedule B 15 mg (N=12) | Oral Arm - Schedule B 20mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 0 | 0 | 0
Anisocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 1 | 5 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 9 | 3 | 5 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 2 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 1 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 2 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 4 | 1 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 8 | 3 | 7 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 14 | 4 | 4 | 2
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 5 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 7 | 3 | 2 | 1
Asthenia (General disorders) | 5 | 4 | 4 | 3 | 1 | 2
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 2 | 3 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 7 | 2 | 5 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 5 | 0 | 1 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 2 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 4 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 3 | 2 | 3 | 0
Thrombosis in device (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Blood amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 1 | 1 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT shortened (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 2 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 8 | 0 | 4 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 1 | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 5 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 10 | 0 | 2 | 0
Headache (Nervous system disorders) | 4 | 6 | 7 | 0 | 5 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Breast discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 7 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 7 | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0
Lividity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 2 | 0 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.